CLINICAL TRIAL: NCT00114660
Title: Topical Application of Cocoa Butter for Prevention of Striae Gravidarum
Brief Title: Cocoa Butter for Prevention of Stretch Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Dr. Fadia Homeidan, American University of Beirut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FM.HO.01; R588416
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Striae Gravidarum; Pregnancy
Keywords: striae gravidarum; stretch marks; cocoa butter; prevention
MeSH Terms: conditions — Striae Distensae

INTERVENTIONS:
Drug: Cocoa butter application

SUMMARY:
This study will check to see if using cocoa butter lotion on the belly, breasts and thighs will help reduce the appearance of stretch marks in pregnancy. Women entering the study will either receive a lotion containing cocoa butter with vitamin E or a lotion containing only vitamin E. After delivery, the study investigators will evaluate whether the women who used cocoa butter lotion were less likely to develop stretch marks.

DETAILED DESCRIPTION:
Primigravid women presenting for prenatal care in the first trimester will be recruited to participate in the study. They will be randomly assigned to receive the study lotion (a commercially available lotion containing cocoa butter with viatmin E), a placebo lotion (a lotion containing vitamin E but no cocoa butter). Participants and investigators will be blinded to the lotion assignment.

Women will be asked to apply a thin layer of the lotion to their abdomen, breasts and thighs once daily until the date of delivery. Participants will be recruited as early in their pregnancy as possible but will not be asked to start applying the lotion before 12 weeks of pregnancy. Women presenting after 20 weeks of pregnancy will not be eligible to participate in the study. The cocoa butter and placebo lotions have been made up to look, smell and feel the same and will be provided to the participants in identical containers. Women who have known hypersensitivity to cocoa butter or any of the components of the lotion will be excluded from the study.

Participants will be assessed at study entry for presence of stretch marks. Baseline information will be collected at that time including pre-pregnancy weight, skin type, and history of stretch marks in the mother or siblings. Women will then be followed up monthly by telephone to assess compliance with the regimen and ensure that they are not developing skin reactions.

Participants will be assessed for the development of stretch marks after delivery. Women will also be asked to provide their own assessment of their skin condition in terms of presence/absence of stretch marks and their severity.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid women in first trimester of pregnancy

Exclusion Criteria:

* Hypersensitivity of cocoa butter

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2004-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Development of stretch marks

CONTACTS AND LOCATIONS:
Overall Officials: Hibah Osman, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Result] Osman H, Usta IM, Rubeiz N, Abu-Rustum R, Charara I, Nassar AH. Cocoa butter lotion for prevention of striae gravidarum: a double-blind, randomised and placebo-controlled trial. BJOG. 2008 Aug;115(9):1138-42. doi: 10.1111/j.1471-0528.2008.01796.x. PMID 18715434